CLINICAL TRIAL: NCT02533999
Title: Assessment of 14-Day Outcomes With the Peak® Surgery System Versus the Traditional Electrocautery Method in Children Ages 3 to 18 Years Undergoing Tonsillectomy With Adenoidectomy for Sleep Disordered Breathing
Brief Title: Peak(R) vs. Electrocautery in Children Undergoing Tonsillectomy With Adenoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Baptist Health Wolfson Children's Hospital (Unknown); Baptist Health Wolfson Surgery Center (Unknown)
Responsible Party: Principal Investigator, Kathryn Blake, PharmD, Director, Center for Pharmacogenomics and Translational Research, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-13
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Electrosurgery

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Instrument (Experimental): PEAK® Plasma Surgery System [PEAK PlasmaBlade® TnA Tonsil and Adenoid Tissue Dissection Device] (Medtronic, Inc) is a marketed device. The PEAK® system generates plasma, "an electrically conductive cloud produced when radiofrequency energy contacting tissue and the tissue breaks down". The system was designed to have the precision of a scalpel, minimal bleeding as with electrosurgery, but reduced collateral thermal tissue damage. The PEAK® Plasma System setting will be standardized for tonsils, to 2 for coagulation and 1 for cutting; and for adenoids, to 7 for coagulation, and 7 for cutting.
  Interventions: Device: PEAK® Plasma System
- Electrosurgery (Active Comparator): Electrosurgery, also known as thermal cautery, refers to a process in which a direct or alternating current is passed through a resistant metal wire electrode, generating heat. The heated electrode is then applied to living tissue to achieve hemostasis or varying degrees of tissue destruction. It is commonly used for tonsillectomy and adenoidectomy in pediatric patients. The electrocautery setting will be standardized to 12 for tonsils and 30 for adenoids.
  Interventions: Device: Electrosurgery

INTERVENTIONS:
Device: PEAK® Plasma System — Surgical method for tonsillectomy and adenoidectomy.
  Arms: Surgical Instrument
Device: Electrosurgery — Surgical method for tonsillectomy and adenoidectomy.
  Arms: Electrosurgery

SUMMARY:
Given the large numbers of children who undergo tonsillectomy (by the time a child is 15 years old, 13% of his/her peers will have had a tonsillectomy), the significant morbidity, and direct and indirect costs associated with absences for child from school or parent from work or other responsibilities, it is vitally important to identify surgical techniques which will minimize pain and serious negative outcomes. This study aims to compare a new surgical technique, PEAK® Surgery System, with electrocautery, one of the most commonly used methods for tonsillectomy with or without adenoidectomy in children 3 to 6 years old with a diagnosis of sleep-disordered breathing.

In this project, the investigator will evaluate intra-operative outcomes including, surgery time and bleeding rates, and post-operative pain scores, bleeding rates, time to resumption of normal diet and activity, analgesic type and use, and frequency of emergent visits over 14 days following surgery.

The hypothesis is that there is no difference in outcomes between the traditional extracapsular electrocautery dissection method of tonsillectomy versus the newly introduced Peak® Surgery System.

The long-term goal is to minimize pain and risk of bleeding and shorten the time to resumption of normal eating and activities in children undergoing tonsillectomy.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

* Specific Aim 1: To assess differences in pain control, assessed by validated pain scores and requirement for postoperative analgesia, during the 14-day post-operative period.
* Specific Aim 2: To assess differences in bleeding (hemorrhage) both intraoperatively and 24 hours post-surgery (immediate period) and between 24 hours and 14 days post-operatively (delayed period).
* Specific Aim 3: To assess differences in other outcomes (time to resumption of normal diet and activities) and adverse events (emergent visits for medical care) between 24 hours and 14 days post-operatively.

BACKGROUND AND SIGNIFICANCE:

Epidemiology of Tonsillectomy in Children. Tonsillectomy is the second most commonly performed procedure in children under 15 years old, second to myringotomy and pressure equalization tube placement. It is estimated that 583,000 outpatient tonsillectomy procedures were performed in children in the US in 2006 accounting for 16% of all ambulatory surgeries with the greatest number (103/10,000) in children ages 0 to 6 years old. In this age group, diagnosis of airway obstruction or sleep disturbance accounts for the majority of surgery indications and tonsillectomy with adenoidectomy account for 90% of the procedures performed (vs. 10% for tonsillectomy alone). Nemours Jacksonville surgeons performed 995 tonsillectomies with/without adenoidectomy at Wolfson Children's Hospital in children 3 to 6 years old with sleep-disordered breathing from 2010-2011.

In this project, the investigators will compare electrocautery surgical method with the PEAK® Plasma Surgery System [PEAK PlasmaBlade® TnA Tonsil and Adenoid Tissue Dissection Device] (Medtronic, Inc), a recently marketed device. There are no published studies comparing the PEAK® system with other traditional methods of performing adenotonsillectomy. Nemours otolaryngologists currently use the PEAK® system for adenotonsillectomies in children 3 to 18 years of age with a diagnosis of sleep-disordered breathing. The PEAK® system generates plasma, "an electrically conductive cloud produced when radiofrequency energy contacting tissue and the tissue breaks down". The system was designed to have the precision of a scalpel, minimal bleeding as with electrosurgery, but reduced collateral thermal tissue damage. Data from the Medtronic website indicates the temperature profile from the PEAK® system to be approximately half that associated electrosurgery at similar cut settings; and human studies indicate a 66% to 80% reduction in thermal injury depth.

PRELIMINARY STUDIES:

There are no preliminary data from Nemours using the Peak® Plasma System.

APPROACH:

1. Study Design This is a prospective, randomized, single-blind controlled study. Patients and caregivers and the study coordinator will be blinded to the surgical method.

This project will involve a single study visit and 6 phone calls and completion of daily diaries for 14 days following surgery and completion of the Glasgow Children's Benefit Inventory 7 6-months after surgery. Parents and caregivers will be contacted after the surgery date is scheduled to discuss the project and determine interest. If interested, and inclusion/exclusion criteria are met, families will be advised of the study and invited to participate. Parental permission will be obtained from the parent/caregiver prior to surgery. Children aged 3 to 18 years old will be included.

Stopping Criteria: The study will be stopped and unblinded if the rate of postoperative hemorrhage, defined as Level II or Level III, exceeds 2 participants in the same surgical group assessed during the first 5-days post-operatively after the first 30 patients have been enrolled. Post-operative bleeding will be defined as follows:

Level I. All children who report to have any history of postoperative hemorrhage, whether or not there is clinical evidence.

Level II. All children who require inpatient admission for postoperative hemorrhage regardless of the need for operative intervention. This level excludes children undergoing evaluation in the emergency department for reported postoperative hemorrhage who have no evidence of clot formation or hemorrhage and are deemed safe for discharge.

Level III. All children who require a return to the operating department for control of postoperative bleeding.

Patients will be instructed to call the clinic if there is more than one tablespoon of blood in a single episode or persistent bleeding of small amounts throughout the day. Administration of dexamethasone perioperatively has been found to not increase the risk of Level II or Level III bleeds in a recent study.

Randomization Children will be randomized in a block design such that an equal number of children are randomized to electrocautery or PEAK® Plasma System for each surgeon. Caregivers will be blinded to surgical technique. The surgeon will have no input into which device a child is randomized. The study coordinator will be blinded as to which device the child was randomized.

Surgical Techniques and Post-Operative Care Surgical Procedure: Patients will be prepped as usual for routine adenotonsillectomy procedure. The procedure will be performed under general anesthesia by a fellowship trained pediatric anesthesiologist. All patients will receive 0.5mg/kg dose of intravenous dexamethasone (maximum 15mg) 11 at the onset of the procedure. Patients requiring adenoidectomy will undergo either curette removal followed by suction electrocautery or ablation by suction electrocautery alone. Adenoidectomy technique will be based upon the size of the adenoid pad where enlarged adenoids routinely employ the curette.

Most children in this age group will receive a premedication of midazolam 0.5 mg/kg prn for anxiety. General anesthesia will be induced by face mask, with sevoflurane, nitrous oxide and oxygen. A peripheral IV will be started and intravenous fentanyl (1-2 ug/kg) will be administered. Propofol may be administered at the discretion of the anesthesiologist. The patient's trachea will be intubated under direct laryngoscopy. The patient will also receive IV dexamethasone, ondansetron, and additional fentanyl, if needed. The maintenance anesthetic will include desflurane, with nitrous oxide and oxygen. At the end of the surgery the patient's trachea will be extubated when the patient is awake. Post-op rescue analgesics will include fentanyl and /or morphine.

Instrument Settings: Settings and methods for electrocautery and the PEAK® Plasma System will be standardized between the surgeons. For the PEAK® Plasma System, the setting will be standardized for tonsils, to 2 for coagulation and 1 for cutting; and for adenoids, to 7 for coagulation, and 7 for cutting. For electrocautery, the setting will be standardized to 12 for tonsils and 30 for adenoids.

Data Collected Intra-operatively Total blood loss will be determined by the method described by Walner, et al in which the operating nurse will record the blood loss based on the amount in the suction canister or suction tubing at the conclusion of each procedure. Data extraction of blood loss from the operative report will be performed by the data entry specialist and not the study coordinator to prevent unblinding of the study coordinator. The Biomedical Research Department has several highly trained data entry specialists who extract clinical data from the EHR.

Data Collected Post-operatively Parents will complete a diary card beginning on the day of surgery and continuing for 14 days. After 30±4 days following surgery, the study coordinator will contact parent of each patient by telephone to obtain information on incidence of late-complications and to collect a global assessment of the parent's perception of the 30-day postoperative period. Assessment will consist of asking parents to state whether their child's pain had been less, the same, or more than they had expected it to be after the adenotonsillectomy. At this assessment, the coordinator and parents will still be blinded to the treatment received. At six-months post-operatively, parents will be mailed the Glasgow Children's Benefit Inventory (GCBI). Unblinding information will be mailed to parents 2 weeks after the GCBI has been mailed.

The following measures will be collected daily on the diary card beginning on Day 0 (day of surgery):

1. Presence of bleeding.

   Post-operative bleeding will be scored as follows:
   * Level I. All children who report to have any history of postoperative hemorrhage, whether or not there is clinical evidence.
   * Level II. All children who require inpatient admission for postoperative hemorrhage regardless of the need for operative intervention. This level excludes children undergoing evaluation in the emergency department for reported postoperative hemorrhage who have no evidence of clot formation or hemorrhage and are deemed safe for discharge.
   * Level III. All children who require a return to the operating department for control of postoperative bleeding.

   Children who return to the emergency department (ED) or hospital who are subsequently diagnosed with Von Willebrand's disease will be excluded from the study and will not be included in the data analysis.
2. Assessment of subjective pain. The child will be asked by the parent to grade severity of pain daily using the Wong-Baker FACES pain rating scale 13 in the morning before eating, drinking, or taking analgesics. The Wong-Baker FACES pain rating scale is a 0 to 10 numerical rating scale (0, 2, 4, 6, 8, 10) with faces indicating the level of pain from a happy face at a score of 0 to a crying face at a score of 10. The scale is recommended for children 3 years and older.
3. Type and frequency of pain medication will be recorded.
4. Return to normal diet. Normal diet is defined as consumption of the types and amount of food such that another family member would not be able to recognize that the patient had undergone throat surgery. Dietary progression from liquid to soft and solid food will be also documented. Diet will be scored as 1, liquids and soft diet only; 2, some solids; 3, mostly solids; and 4, normal diet.
5. Return to normal activity. Normal activity is defined as carrying out the same types and amounts of daily activity as before surgery, even if still associated with fatigue. Activity will be scored as 1, none; 2, very little; 3, mostly normal; 4, normal.
6. At each post-operative phone call, the study coordinator will collect data regarding bleeding events with the questions below and document parental phone calls or visits to physician regarding parental concerns over child's recovery.

Data Collected After 6-Months Six months following surgery, parents will be mailed the Glasgow Children's Benefit Inventory (GCBI) 7. The GCBI is a post intervention health-related benefit measure consisting of 24 broadly worded yes/no questions that are applicable to any area of pediatric medicine. The GCBI scores will be compared between surgical techniques. The two study groups will be matched for age and sex.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are aged 3 up to 18 years old; children younger than 3 years are excluded because of a higher risk of perioperative complications such as requiring an overnight hospitalization and dehydration after discharge resulting in an emergency department visit or hospitalization
2. Clinical diagnosis of sleep disordered breathing or obstructive sleep apnea 10 or recurrent tonsillitis
3. Presence of adenotonsillar hypertrophy

Exclusion Criteria:

1. Diagnosis of bleeding disorders*
2. Craniofacial malformation
3. Previous adenotonsillectomy
4. Suspected lymphoma
5. Developmental delay
6. Diabetes or any other disease that slows wound healing
7. Peritonsillar abscess
8. Expressive language disorder
9. Hematologic wound healing disorder or necrotizing dermatosis,
10. Implanted electric device
11. Mucopolysaccharidosis
12. Use of nonsteroidal anti-inflammatory drugs in the two weeks prior to the surgery
13. Allergy to medication(s) used in this protocol
14. Other planned surgical procedure during this surgical period
15. Chronic pain disorder
16. Planned hospital admission

    * We will use the following set of questions to evaluate for bleeding issues. If all are answered "no", then the child will be enrolled. If any are answered "yes", the child will be excluded and the family will be referred for a Hematology consult.

      1. Has your child been told he/she has a bleeding disorder?
      2. Does anyone in the child's family (grandmother, grandfather, mother, father, siblings) have a known bleeding disorder?
      3. Does your child have easy bruising or difficulty stopping bleeding when he/she gets a cut or scratch?
      4. If your child has had had surgery before, did the surgeon indicate that controlling bleeding was difficult or was your child required to come back to the hospital for bleeding control?

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Blake, PharmD, Principal Investigator — Nemours Children's Specialty Care

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surgical Instrument | Electrosurgery
Started | 38 | 37
Completed | 32 | 30
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 3 | 5
Not completed — Protocol Violation | 3 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Randomized but intervention not received | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgical Instrument | Electrosurgery | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32 | 30 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62

OUTCOME MEASURES:

1. Primary Outcome: Pain Control Assessed by Validated Pain Scores: Days to Having no Pain Following Surgery
Description: To assess differences in pain control, assessed by validated pain scores and requirement for postoperative analgesia, during the 14-day post-operative period in children ages 3 to 18 years undergoing adenotonsillectomy with a clinical diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
  Assessment of subjective pain. The child will be asked by the parent to grade severity of pain daily using the Wong-Baker FACES pain rating scale in the morning before eating, drinking, or taking analgesics. The Wong-Baker FACES pain rating scale is a 0 to 10 numerical rating scale (0, 2, 4, 6, 8, 10) with faces indicating the level of pain from a happy face at a score of 0 to a crying face at a score of 10. The scale is recommended for children 3 years and older.
  Type and frequency of pain medication will be recorded.
Time Frame: during the 14-day post-operative period
Population: Patients aged 3- to 17-years scheduled for adenotonsillectomy with a clinical diagnosis of sleep disordered breathing, or obstructive sleep apnea with adenotonsillar hypertrophy, or recurrent adenotonsillitis were enrolled between October 2013 and June 2015.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Days | 7.0 [5.2 to 8.6] | 9.0 [8.0 to 10.0]

2. Secondary Outcome: Number of Participants Who Experienced Bleeding Intraoperatively and 24 Hours Post-surgery (Primary Period)
Description: To assess differences in bleeding (hemorrhage) rate (either Level I, Level II, or Level III) intraoperatively and 24 hours post-surgery (primary period) in children ages 3 to 18 years undergoing adenotonsillectomy with a diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
  Post-operative bleeding will be scored as follows:
  Level I. All children who report to have any history of postoperative hemorrhage, whether or not there is clinical evidence.
  Level II. All children who require inpatient admission for postoperative hemorrhage regardless of the need for operative intervention.
  Level III. All children who require a return to the operating department for control of postoperative bleeding.
Time Frame: intraoperatively and 24 hours post-surgery (primary period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Participants | 0 | 0

3. Secondary Outcome: Number of Participants Who Experienced Bleeding Between 24 Hours and 14 Days Post-operatively (Secondary Period)
Description: To assess differences in bleeding (hemorrhage) rate (either Level I, Level II, or Level III) between 24 hours and 14 days post-operatively (secondary period) in children ages 3 to 18 years undergoing adenotonsillectomy with a diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
  Post-operative bleeding will be scored as follows:
  Level I. All children who report to have any history of postoperative hemorrhage, whether or not there is clinical evidence.
  Level II. All children who require inpatient admission for postoperative hemorrhage regardless of the need for operative intervention. Level III. All children who require a return to the operating department for control of postoperative bleeding.
Time Frame: between 24 hours and 14 days post-operatively (secondary period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Participants | 0 | 1

4. Secondary Outcome: Days to Resumption of Normal Diet
Description: To assess differences in other outcomes (time to resumption of normal diet) from discharge to 14 days post-operatively in children ages 3 to 18 years undergoing adenotonsillectomy with a diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
  Return to normal diet. Normal diet is defined as consumption of the types and amount of food such that another family member would not be able to recognize that the patient had undergone throat surgery. Dietary progression from liquid to soft and solid food will be also documented. Diet will be scored as 1, liquids and soft diet only; 2, some solids; 3, mostly solids; and 4, normal diet.
Time Frame: from discharge to 14 days post-operatively
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Days | 9.0 [6.4 to 11.6] | 8.0 [5.7 to 10.3]

5. Secondary Outcome: Days to Resumption of Normal Activities
Description: To assess differences in other outcomes (time to resumption of normal activities) from discharge to 14 days post-operatively in children ages 3 to 18 years undergoing adenotonsillectomy with a diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
  Return to normal activity. Normal activity is defined as carrying out the same types and amounts of daily activity as before surgery, even if still associated with fatigue. Activity will be scored as 1, none; 2, very little; 3, mostly normal; 4, normal.
Time Frame: from discharge to 14 days post-operatively
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Days | 7.0 [6.2 to 7.8] | 8.0 [5.8 to 8.2]

6. Secondary Outcome: Adverse Events (Emergent Visits for Medical Care)
Description: To assess differences in adverse events (emergent visits for medical care) from discharge to 14 days post-operatively in children ages 3 to 18 years undergoing adenotonsillectomy with a diagnosis of sleep-disordered breathing using the traditional Extracapsular Electrocautery Dissection Method versus the Peak® Surgery System Method.
Time Frame: from discharge to 14 days post-operatively
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
Participants | 2 | 1

7. Other Pre Specified Outcome: Glasgow Children's Benefit Inventory (GCBI)
Description: A composite score of GCBI for each patient will be calculated by assigning the individual question responses a numerical value from -2 to +2, then adding these up, dividing by the number of questions (24), and multiplying by 50 to produce a result on a scale from -100 (maximum harm) to+ 100 (maximum benefit) .
Time Frame: At six-months post-operatively
Population: as for outcome 1
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Surgical Instrument | Electrosurgery
Number analyzed (Participants) | 32 | 30
scores on a scale | 34.8 (4.6) | 29.1 (4.2)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a 30-day period following surgery.
Description: The clinicaltrials.gov definitions were used. Participants were queried regarding any adverse events at each follow up phone call during the 14-day post operative period and at the 30-day post operative phone call.
Arm/Group | Surgical Instrument | Electrosurgery
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/30
Other Adverse Events (participants affected / at risk) | 2/32 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Instrument (N=32) | Electrosurgery (N=30)
Tonsilar bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Tonsilar bleeding (Level II) resulting in hospitalization overnight.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Instrument (N=32) | Electrosurgery (N=30)
Fever (General disorders) | 2 (2) | 0 (0) — Visit to emergency department due to dehydration (fever and dehydration occurred together in the 2 participants reported).
Dehydration (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Visit to emergency department due to dehydration (fever and dehydration occurred together in the 2 participants reported).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No